CLINICAL TRIAL: NCT02622594
Title: A Randomized, Evaluator-blinded, Bilateral Comparison of the Treatment of Facial Actinic Keratoses Using Combination Microneedling and Photodynamic Therapy With Aminolevulinic Acid and Blue Light Versus Photodynamic Therapy With Aminolevulinic Acid and Blue Light Using Two Different Incubation Times
Brief Title: Bilateral Comparison of Treatment of Facial Actinic Keratoses Using Microneedling and Photodynamic Therapy With Aminolevulinic Acid and Blue Light Versus Photodynamic Therapy With Aminolevulinic Acid and Blue Light Using Two Incubation Times
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dermatology, Laser & Vein Specialists of the Carolinas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADV Microneedling/PDT 002; NCT02579447 (obsolete NCT alias)
Record Dates: First submitted 2015-10-22; First posted 2015-12-04 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Treatment 1 will include microneedling performed prior to ALA application to their right face and ALA application only to the left face 60 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds).
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: Environ Cosmetic Roller; Device: BLU-U IIlluminator
- 2 (Active Comparator): Treatment 2 will include microneedling performed prior to ALA application to their left face and ALA application only to the right side of their face 60 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds).
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: Environ Cosmetic Roller; Device: BLU-U IIlluminator
- 3 (Active Comparator): Treatment 3 will include microneedling performed prior to ALA application to their right face and ALA application only to the left side of their face 30 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds).
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: Environ Cosmetic Roller; Device: BLU-U IIlluminator
- 4 (Active Comparator): Treatment 4 will include microneedling performed prior to ALA application to their left face and ALA application only to the right side of their face 30 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds).
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: Environ Cosmetic Roller; Device: BLU-U IIlluminator

INTERVENTIONS:
Drug: Aminolevulinic Acid (ALA)
  Other Names: Levulan Kerastick applicator
Device: Environ Cosmetic Roller
  Other Names: Microneeling
Device: BLU-U IIlluminator
  Other Names: Blue light

SUMMARY:
This is an investigator initiated, two center, randomized, evaluator-blinded, bilateral (right vs. left) study of photodynamic therapy in subjects with facial actinic keratoses.

Subject's face will be randomized to receive one of four treatments: Treatment 1, Treatment 2, Treatment 3 or Treatment 4. Treatment 1 will include microneedling performed prior to ALA application to their right face and ALA application only to the left face 60 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds). Treatment 2 will include microneedling performed prior to ALA application to their left face and ALA application only to the right side of their face 60 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds). Treatment 3 will include microneedling performed prior to ALA application to their right face and ALA application only to the left side of their face 30 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds). Treatment 4 will include microneedling performed prior to ALA application to their left face and ALA application only to the right side of their face 30 minutes prior to BLUE light treatment for 1000 seconds (16 minutes 40 seconds). The face is defined as the surface of the skin encompassing the forehead to the hair line and tops of the eyebrows, the entire nasal dorsum, the cheeks (bounded by the orbital rim, the anterior border of the ear, the jawline, the nose and the chin), the upper lip (not including the vermilion border) and the chin (bounded by the lower edge of the vermilion border, the cheek junction and the jawline). The treatment areas will be not be occluded. A line will be drawn with a marker that intersects the nose, forehead, upper lip and chin in the midline. The left face is defined as the face to the left of this line and the right face is defined as the face to the right of this line. Posttreatment follow-up visits will be scheduled to occur 48 hours after the treatment and at 1, 3 and 6 months after the treatment. A blinded evaluator who will remain blinded with respect to the randomization will conduct grading of the subject's actinic keratoses and photodamage. Tolerability of treatment will be assessed by evaluations of the local skin response (erythema, edema, etc.) and will be conducted by an unblinded evaluator.

Safety will be evaluated by adverse events and local skin responses reported during the study

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female over the age of 18 years. Females must be post-menopausal, surgically sterile or using a medically acceptable form of birth control, with a negative urine pregnancy test at the Baseline visit.
* Subject has provided written and verbal informed consent.
* Subject has four (4) or more AK lesions on each side of the face.
* Subject is willing to comply with study instructions and return to the clinic for required visits.
* Subject has Fitzpatrick skin type I-IV

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has a history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis or any condition with associated immunosuppression (e.g. HIV, systemic malignancy, etc.).
* Subject has any skin pathology or condition that could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy.
* Subject has any condition, which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
* Subject has Fitzpatrick skin type V - VI.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment (baseline).
* Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
* Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.
* Subject has a known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol).
* Subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
* Subject has used any of the following topical preparations on the area(s) to be treated
* Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g. glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment.
* Retinoids, including tazarotene, adapalene, tretinoin, retinol, within 4 weeks of the initiation of treatment.
* Cryotherapy, dicofenac or other treatments for AK within 8 weeks of initiation of treatment
* Microdermabrasion, laser ablative treatments or chemical peels within 8 weeks of the initiation of treatment.
* 5-FU, imiquimod or ALA-PDT within 6 months of initiation of treatment.
* Subject has used any of the following systemic medications:
* Immuno-suppressants including steroids, chemotherapy, etc. within 3 months of the initiation of treatment
* Retinoid therapy within 6 months of the initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Efficacy-Percentage of treatment areas with >75% reduction in lesion count as compared to baseline | 6 months
Efficacy-Percentage of treatment areas with 100% cure rate as compared to baseline | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina, United States